CLINICAL TRIAL: NCT05437666
Title: Effects of Pelvic Floor Health Education Program in Women With Stress Urinary Incontinence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, seyda toprak celenay, associate professor, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022/06/27
Record Dates: First submitted 2022-06-27; First posted 2022-06-29 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Educational Status

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education group (Experimental): The education program was given both an educational presentation and a booklet related to the pelvic floor health
  Interventions: Other: Education and booklet
- Control group (Other): The control group will be given a booklet related to the pelvic floor health
  Interventions: Other: Booklet

INTERVENTIONS:
Other: Education and booklet — The education program was given both an educational presentation accompanied by a physiotherapist once a week for six weeks and a booklet related to the pelvic floor health (pelvic floor, urinary incontinence, risk factors, treatment options, healthy behavioral strategies etc.)
  Arms: Education group
Other: Booklet — The control group will be given a booklet related to the pelvic floor health (pelvic floor, urinary incontinence, risk factors, treatment options, healthy behavioral strategies etc.)
  Arms: Control group

SUMMARY:
The aim of this study is to investigate the effects of pelvic floor health education program on urinary incontinence symptoms, knowledge level and quality of life in women with stress urinary incontinence.

DETAILED DESCRIPTION:
Stress urinary incontinence (SUI) is the involuntary urinary incontinence that develops in parallel with the increase in intra-abdominal pressure and is seen in the absence of detrusor contraction. Studies have shown that SUI, leading to a decrease in the quality of life and worsening of social and health conditions, is more common in women than men.

Knowledge of pelvic floor health or urinary incontinence is generally low. Low level of knowledge or wrong information limits patients' access to treatment. Pelvic floor muscle exercise and lifestyle recommendations are also the first treatment options for SUI.

The information and awareness related to the pelvic floor and SUI can be increase and unhealthy behavioral strategies can be modifiable through education programs. Therefore the education programs related to the pelvic floor health would have positive effects on urinary incontinence symptoms, knowledge level and quality of life. Studies about this issue are needed.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65
* Women with stress urinary incontinence
* Those who volunteered to participate in the study
* Being literate

Exclusion Criteria:

* Having advanced pelvic organ prolapse
* Having a malignancy
* Having a urinary tract infection
* Those who have a problem that interferes with cooperation and understanding

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women with stress urinary incontinence
Enrollment: 40 (Estimated)
Dates: Start 2022-07-15 (Estimated); Primary Completion 2022-10-15 (Estimated); Study Completion 2023-07-15 (Estimated)

PRIMARY OUTCOMES:
Presence of urinary incontinence symptoms | change from baseline at 6 weeks
  International Consultation on Incontinence Questionnaire-Short Form will be used to evaluate the urinary incontinence symptoms. The scale has 6 questions and 4 dimensions (frequency, severity, type of urinary incontinence, and its effect on daily life). The score to be obtained from the scale varies between "0" and "21". As the score increases, the urinary incontinence symptoms also increases.

SECONDARY OUTCOMES:
Pelvic floor health knowledge level | change from baseline at 6 weeks
  Pelvic Floor Health Knowledge Quiz will be used to evaluate the knowledge level of patients about general pelvic floor health. It consists of 3 subscales (function/dysfunction, risk/etiology subscale and diagnosing/treatment) and total 29 questions.
  Total score is calculated by summing the number of correct responses, which range between 0 and 29, where a higher score indicates a higher level of knowledge about the pelvic floor health
Urinary incontinence konwledge level | change from baseline at 6 weeks
  The Prolapse Incontinence Knowledge Quiz-urinary incontinence subscale will be used to evaluate the knowledge level of the urinary incontinence. It consists of 12 items. Total score is calculated by summing the number of correct responses, which range between 0 and 12, where a higher score indicates a higher level of knowledge about urinary incontinence.
Life quality | change from baseline at 6 weeks
  King Health Questionnaire will be used to evaluate the life quality. The questionnaire, consisting of thirty-two items, consists of 2 parts. In the first part, there are 2 questions questioning the general health perception and incontinence effect, and 19 questions dividing the quality of life into 7 areas (role limitations, physical limitations, social limitations, personal relationships, emotional problems, sleep/energy disorders, symptom severity measurement). In the second part, there are 11-item complaint severity scales that evaluate the presence and severity of urinary symptoms. While the best score that can be obtained on the complaint severity scale is "0", the worst score is "30", the best score that can be obtained for all King Health Questionnaire subsections is "0" and the worst score is "100".
Compliance with the program | after program (6th week)
  Compliance with the program will be evaluated using a 10-cm visual analog scale. 0 point indicates "did not comply with the program" and 10 point indicates " complied with the program".

CONTACTS AND LOCATIONS:
Overall Officials: Seyda Toprak Celenay, Principal Investigator — Ankara Yildirim Beyazıt University